CLINICAL TRIAL: NCT06065020
Title: Pilot Trial of an Evidence-based Community Intervention to Improve Depressive Symptoms Among Peruvian Older Adults
Brief Title: Community Intervention to Improve Depressive Symptoms Among Older Adults (VIDACTIVA)
Acronym: VIDACTIVA1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de San Martín de Porres (Other)
Collaborators: Asociacion Benefica Prisma (Other); Johns Hopkins University (Other); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E10012021018
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-08

CONDITIONS: Depression, Anxiety
Keywords: depression; aged; problem-solving
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Standard of Care

STUDY DESIGN:
Masking Description: We will try to mask the outcome assessor, but for the nature of the intervention, it will be difficult that outcome assessor remain blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): VIDACTIVA program
  Interventions: Behavioral: VIDACTIVA sessions
- Control group (Active Comparator): Standard Care
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: VIDACTIVA sessions — Community health workers (CHWs) will delivered VIDACTIVA intervention that consists in 8 home-sessions, one hour duration, within a period of 14 weeks + 2 follow-up calls (monthly). In total, a period of 22 weeks.
  The multicomponent intervention consist in the following:
  Problem-Solving Exercises: These are basic structured exercises aimed at training older individuals in problem-solving. This activity is centered around the older adult, meaning the older adults guides this activity, and the CHWs is a facilitator.
  Physical Activation: This component involves planning and "scheduling" enjoyable activities (physical or social) that the older adult chooses based on their preferences and capabilities.
  Education on Depressive Symptoms (psychoeducation)
  Arms: Intervention group
Behavioral: Standard Care — Study fieldworkers will provide 2 educational sessions (45-60 min) about mental health at old age and participant will be guided to mental health community services (primary care centers). One session after the enrolment (week 1) and one at the 14th week.
  Arms: Control group

SUMMARY:
The goal of this pilot trial is to test how feasible is to conduct a large clinical trial that evaluate both implementation and effectiveness outcomes of a community-based interventions for older adults with depression in low-resource urban settings from Lima, Peru.

The main questions:

Is the way we are planning the study, including those who are taking part and what they will do, good for a large study?

Is the interventional package we are developing good the way it is, and can it be done the way we planned it?

DETAILED DESCRIPTION:
Participants who join will be split into two groups: one group will get the interventional program, and the other group will get standard care. In the interventional group, community health workers will meet with participants eight times to do activities and talk about how they feel. The standard group will have two visits where they will learn things about mental health.

The results of the study will help the researchers understand whether they can test the program in larger study. Additionally, see whether those participants in the interventional group feel better than those who are in the standard group.

Sample size: This is a pilot trial. No sample size calculations are needed because the objective is NOT to evaluate the effect of the intervention, but rather the feasibility of conducting a large-scale clinical trial. It is expected to enroll 64 participants (32 control group vs 32 intervention group). This number is based on previous formative study and training of community health workers.

Researchers will collect basic information to assess feasibility for a larger trial, including:

* Number of potential participants screened per month;
* Number of participants enroled per month;
* Average time from enrolment to randomisation.
* Average time to reach enrolment goal
* Proportion of eligible participants who enrol
* Proportion of people who maintain the study in both groups.
* Reasons for abandoning the study.
* Visit durations

ELIGIBILITY:
Inclusion Criteria:

* Having depressive symptoms (score equal to or greater than 6 on the Patient Health Questionnaire - PHQ 9).
* Capacity to give consent.
* Current residence in Villa El Salvador, Lima, Peru.

Exclusion Criteria:

* Previous diagnosis of bipolar disorder
* History of substance abuse
* History of dissociative disorder, psychosis or dementia, or moderate memory and/or cognition problems.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | At baseline, at 14th and 22th week.
  Measured by Patient Health Questionnaire - 9 (PHQ-9) [ minimum score: 0 ; maximum score: 27 ] [More score = worse symptoms]

SECONDARY OUTCOMES:
Anxiety symptoms | At baseline, at 14th and 22th week.
  Measured by Generalised Anxiety Disorder - 7 (GAD-7) [min score: 0 , max score: 21] [more score, worse symptoms]
Loneliness | At baseline, at 14th and 22th week.
  Measured by the Three-Items Loneliness [min 0, max: 9] [more score, more lonely]

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Flores-Flores, MD, MSc, Principal Investigator — Universidad de San Martin de Porres
Locations (1):
- Universidad de San Martin de Porres, Lima, Lima Province, Peru

IPD SHARING:
Plan to Share IPD: Yes
Once first manuscript using data is published.
Supporting Information: Study Protocol, ICF
Time Frame: Expected to be available, once first manuscript is published. Expected 2025. For the next five years (2030).
Access Criteria: We will share data based on reasonable request of a researcher.

REFERENCES:
- [Derived] Otero-Oyague D, Lastra D, Patino V, Carrion I, Cruz-Riquelme T, Pollard SL, Parodi JF, Steinman L, Gallo JJ, Valle R, Castro N, Flores-Flores O. Community health workers fostering trust and engagement in a community-based intervention for depressive older adults in Peru: a qualitative study. Res Sq [Preprint]. 2025 Oct 19:rs.3.rs-7665993. doi: 10.21203/rs.3.rs-7665993/v1. PMID 41282139
- [Derived] Cruz-Riquelme T, Zevallos-Morales A, Carrion I, Otero-Oyague D, Patino V, Lastra D, Valle R, Parodi JF, Pollard SL, Steinman L, Gallo JJ, Flores-Flores O. Pilot trial protocol: community intervention to improve depressive symptoms among Peruvian older adults. Pilot Feasibility Stud. 2024 Aug 22;10(1):112. doi: 10.1186/s40814-024-01540-1. PMID 39175082